CLINICAL TRIAL: NCT06977685
Title: Effect of Non-Selective Beta-Blockers on Outcomes in Patients Discharged After Hospitalization for Acute Decompensation of Cirrhosis: A Retrospective Cohort Study Using Target Trial Emulation Design
Brief Title: Effect of Non-Selective Beta-Blockers on Outcomes in Cirrhosis Patients After Hospitalization: A Retrospective Cohort Using Target Trial Design
Status: Active, not recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: SamsungMC_LC_NSBB_2025
Record Dates: First submitted 2025-05-08; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Cirrhosis; Decompensated Cirrhosis of Liver
Keywords: Non-Selective Beta-Blockers; Decompensated Cirrhosis; Target Trial Emulation
MeSH Terms: conditions — Fibrosis | interventions — Carvedilol; Propranolol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With NSBB: Patients with chronic hepatitis B or C who were hospitalized for hepatic complications (hepatic encephalopathy, hepatorenal syndrome, ascites, or spontaneous peritonitis) and received NSBB prescription at discharge. The study will compare outcomes in this group with the non-NSBB group.
  Interventions: Drug: Non-selective beta-blockers
- Without NSBB: Patients with chronic hepatitis B or C who were hospitalized for hepatic complications (hepatic encephalopathy, hepatorenal syndrome, ascites, or spontaneous peritonitis) and did not receive NSBB prescription at discharge. This group will serve as the control group for comparison.

INTERVENTIONS:
Drug: Non-selective beta-blockers — Non-selective beta-blockers (NSBB) prescribed at discharge for patients hospitalized with hepatic complications. The study will analyze two types of NSBB: propranolol and carvedilol. The study will also examine potential dosage effects by categorizing NSBB use into low-dose and middle-high dose groups. NSBB use is defined as a prescription for at least 2 days at discharge.
  Other Names: Carvedilol; Propranolol
  Groups: With NSBB

SUMMARY:
The goal of this observational study is to learn if non-selective beta-blockers (NSBB) improve outcomes in patients with chronic hepatitis B or C who are discharged after hospitalization for acute decompensation of cirrhosis. The main questions it aims to answer are:

1. Does NSBB use at discharge reduce mortality rates in cirrhotic patients with hepatic complications?
2. Does NSBB use at discharge decrease hospital readmission rates?

Researchers will compare patients discharged with NSBB prescriptions to those without NSBB to see if NSBB use decreases mortality and readmission rates.

Participants were patients hospitalized for hepatic complications (hepatic encephalopathy, hepatorenal syndrome, ascites, or spontaneous peritonitis) between January 2013 and October 2023, with data analyzed retrospectively using a target trial emulation design.

DETAILED DESCRIPTION:
This retrospective cohort study aims to investigate the effects of non-selective beta-blockers (NSBB) on clinical outcomes in patients with chronic hepatitis B or C who were hospitalized for acute decompensation of cirrhosis. The study employs a target trial emulation design to simulate a randomized controlled trial using observational data.

Background and Rationale:

Non-selective beta-blockers are commonly used in patients with cirrhosis to reduce portal pressure and prevent complications. However, their role in patients discharged after hospitalization for hepatic complications remains unclear.

Study Design:

The study uses national health insurance claims data from South Korea to identify eligible patients and their outcomes. To address potential confounding inherent in observational studies, three analytical approaches are employed:

1. Traditional multivariable regression analysis
2. Propensity score matching
3. Inverse probability of treatment weighting (IPTW)

Treatment Definition:

NSBB use is defined as a prescription for at least 2 days at discharge. Two types of NSBB are examined: propranolol and carvedilol. Dosage effects are also explored by categorizing NSBB use into low-dose and middle-high dose groups.

Endpoints:

The primary endpoint is all-cause mortality, while secondary endpoints include all-cause hospital readmission and hepatic complication-related hospital readmission. All endpoints are assessed at 1 month, 3 months, 6 months, and 1 year after discharge.

Statistical Analysis:

Kaplan-Meier survival analyses and Cox proportional hazards models will be used to compare outcomes between treatment groups. Models will be adjusted for demographic factors, comorbidities, concurrent medications, health behaviors, and admission-related variables. Subgroup analyses will be conducted based on age, sex, and type of hepatic complication.

This study aims to provide clinicians with evidence regarding the use of NSBB in patients with viral hepatitis-related cirrhosis following hospitalization for acute decompensation, potentially informing clinical decision-making for this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with liver cirrhosis and chronic hepatitis B or C
* Hospitalized due to hepatic complications (hepatic encephalopathy, hepatorenal syndrome, ascites, or spontaneous peritonitis) between January 2013 and October 2023
* Age 19 years and older

Exclusion Criteria:

* History of bradycardia
* History of hypotension
* History of asthma
* History of cancer
* History of heart failure
* History of myocardial infarction
* History of stroke
* History of chronic kidney disease
* History of chronic obstructive pulmonary disease (COPD)
* History of ischemic heart disease
* Esophageal variceal bleeding during index hospitalization

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include adult patients with liver cirrhosis and chronic hepatitis B or C who were hospitalized due to hepatic complications in South Korea between January 2013 and October 2023. The study will focus on patients who experienced hepatic complications including ascites, peritonitis, hepatorenal syndrome, and hepatic encephalopathy. Both patients who received NSBB at discharge and those who did not will be included in the analysis to allow for comparison between these groups.
Sampling Method: Non-Probability Sample
Enrollment: 7725 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 1 month, 3 months, 6 months, and 1 year after discharge from index hospitalization
  Death from any cause following discharge after hospitalization for hepatic complications of cirrhosis. Mortality data will be obtained through death registry linkage. Hazard ratios (HR) will be calculated using Cox proportional hazards models, adjusted for demographic factors, comorbidities, medications at discharge, health behaviors, and admission-related variables.

SECONDARY OUTCOMES:
All-cause hospital readmission | 1 month, 3 months, 6 months, and 1 year after discharge from index hospitalization
  Any hospital readmission following discharge after the index hospitalization for hepatic complications of cirrhosis. Readmission data will be obtained from hospitalization claims. Hazard ratios (HR) will be calculated using Cox proportional hazards models, adjusted for demographic factors, comorbidities, medications at discharge, health behaviors, and admission-related variables.
Hepatic complication-related hospital readmission | 1 month, 3 months, 6 months, and 1 year after discharge from index hospitalization
  Hospital readmission specifically related to hepatic complications (hepatic encephalopathy, hepatorenal syndrome, ascites, or spontaneous peritonitis) following discharge after the index hospitalization. Readmission data will be categorized based on diagnosis codes in hospitalization claims. The same statistical methods as for all-cause readmission will be applied.

CONTACTS AND LOCATIONS:
Overall Officials: Dong Hyun Sinn, MD, PhD, Principal Investigator — Samsung Medical Center, Sungkyunkwan University School of Medicine
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the sensitive nature of the medical information and patient privacy concerns.